CLINICAL TRIAL: NCT01281930
Title: Abscess Packing Versus Wick Placement After Incision and Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0719 -201103241
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Superficial Abscess Packing
Keywords: Superficial abscess; packing material; wick; incision and drainage
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Wick placement into abscess cavity (Experimental)
  Interventions: Procedure: Wick placement into abscess cavity
- Full packing of abscess cavity (Active Comparator)
  Interventions: Procedure: Full packing into abscess cavity

INTERVENTIONS:
Procedure: Full packing into abscess cavity — After incision and drainage plain 1/4-1/2 inch gauze packing material is placed into the cavity to fill it
  Arms: Full packing of abscess cavity
Procedure: Wick placement into abscess cavity — After incision and drainage of the abscess a piece of plain gauze 1/4-1 inch packing material that is as wide as can be easily passed through the opening is placed into the cavity spanning one diameter of the cavity
  Arms: Wick placement into abscess cavity

SUMMARY:
Abscesses or "boils" are becoming more common every year and are a common reason children come to the Emergency Department. For the abscess to heal the skin needs to be opened to let the pus come out. Often doctors put something called "packing material" or gauze into the abscess space to help aid in healing. It is not known if the type of "packing" that is done is necessary or if a more simple treatment is as good or better. With informed consent we randomly place a child into one (1) of two (2) groups in this study that will say if the child's abscess/boil is packed with gauze in the traditional way or if a wick (small piece) of gauze is placed after the abscess/boil is opened and the fluid is drained. After treatment in the emergency department the child will be scheduled to follow-up in the Pediatric Acute Wound Service (PAWS) clinic as all other children with this infection are scheduled. At this visit the healing of the wound will be checked by the staff in the clinic and will be scored. With this evaluation of the wound the hypothesis that for a simple superficial (skin) abscess/boil a gauze wick placement into the abscess/boil is as effective as placement of traditional gauze packing.

ELIGIBILITY:
Inclusion Criteria:

* Well appearing patient
* Abscesses restricted to the superficial areas of the extremities, buttocks, abdominal and thoracic walls, and back
* Patients presenting Saturday-Wednesday

Exclusion Criteria:

* Fever >38 degrees celsius
* Ill appearing patient
* Underlying immunodeficiency or disorder leading to chronic abscess formation
* Any reason for admission to hospital beyond the need for sedation at the time of follow-up
* Thursday-Friday

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2009-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Abscess healing based upon clinical criteria and clinical judgement | 24-72 hours
  Abscesses are assessed for pus accumulation, erythema from the wound, if the patient has a fever and the overall clinical judgment of the evaluating health care professional at the time of follow-up.

SECONDARY OUTCOMES:
Pain since abscess drainage | 24-72 hours
Parent/guardian comfort with removing the packing material or wick from the abscess cavity | 24-72 hours
Parent/guardian assessment of the abscess wound at 2 weeks | 2 weeks
Parent/guardian assessment of pus drainage at 2 weeks | 2 weeks
Need for further treatment of same abscess within 2 weeks | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States